CLINICAL TRIAL: NCT06396429
Title: Efficacy and Safety of HRS9531 in Overweight or Obese Participants: A Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: To Compare the Efficacy and Safety of HRS9531 and Placebo in Subjects With Overweight or Obese
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9531-301
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A: HRS9531 injection (Experimental)
  Interventions: Drug: HRS9531 injection
- Treatment group B: HRS9531 injection (Experimental)
  Interventions: Drug: HRS9531 injection
- Treatment group C: HRS9531 injection (Experimental)
  Interventions: Drug: HRS9531 injection
- Placebo injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HRS9531 injection — HRS9531 injection; low dose
  Arms: Treatment group A: HRS9531 injection
Drug: HRS9531 injection — HRS9531 injection; medium dose
  Arms: Treatment group B: HRS9531 injection
Drug: HRS9531 injection — HRS9531 injection, high dose
  Arms: Treatment group C: HRS9531 injection
Drug: Placebo — blank preparation, participants received matching placebo.
  Arms: Placebo injection

SUMMARY:
The study aims to evaluate the efficacy and safety of HRS9531 in subjects with overweight or obese for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Male or female subjects, ≥18 years of age at the time of signing informed consent.
3. At screening visit, BMI≥28.0 Kg/m2, or ≥24 Kg/m2 with at least one weight-related complication, such as prediabetes, hypertension, dyslipidemia, obstructive sleep apnea, and nonalcoholic fatty liver disease.
4. Diet and exercise control for at least 3 months before screening visit, and less than 5 kg self-reported change within the last 3 months.
5. Fertile male and female subjects (including partners) have no plans to have children and agree to use effective contraception within 2 months after signing the informed consent form and the last medication, and fertile female or male subjects have no plans to donate eggs/sperm; Fertile female subjects tested negative for regnancy within the first 3 days of randomization and were not lactating.

Exclusion Criteria:

1. Presence of clinically significant lab results at screening visit;
2. Uncontrollable hypertension;
3. PHQ-9 score ≥15;
4. Medical history or illness that affects your weight;
5. History of diabetes;
6. Acute infection, acute trauma, or medium to large surgery within 1 month prior to screening;
7. History of acute cardiovascular and cerebrovascular diseases within 6 months prior to screening;
8. Any organ-system malignancies developed within 5 years except for cured local basal cell cancer of the skin、 in-situ cancer of the cervix and in-situ cancer of the prostate;
9. Confirmed or suspected depression, bipolar disorder, suicidal tendencies, schizophrenia, or other serious mental illness;
10. Known or suspected history of alcohol and/or substance abuse or drug abuse;
11. History of acute or chronic hepatitis or other serious liver disease other than alcoholic fatty liver disease.
12. Have received or plan to have an organ or bone marrow transplant during the study.
13. The presence of any blood disorders that may interfere with HbA1c testing.
14. Autoimmune disease is present and systemic glucocorticoid therapy or immunosuppressive therapy is planned during the study.
15. Use of drugs or treatments that may have caused significant weight gain or loss within the 3 months prior to screening;
16. Weight loss surgery or endoscopic and/or medical device-based weight loss therapy is planned for or during the study period;
17. Use of drugs or treatments that may have caused significant weight gain or loss within the 3 months prior to screening;
18. Patients with blood donation or blood loss ≥400 mL or receiving blood transfusion within 3 months before screening.
19. Surgery is planned during the tria;
20. Mentally incapacitated or speech-impaired subjects are unable to fully understand or participate in the test process；
21. In the investigator's judgment, there are circumstances (medical, psychological, social, or geographical factors, etc.) that affect subject safety or any other conditions that interfere with the evaluation of the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in weight after 48 weeks of treatment | Baseline, Week 48
Proportion of subjects with weight loss of≥5% from baseline after 48 weeks of treatment | Week 48

SECONDARY OUTCOMES:
Proportion of subjects with weight loss of ≥10% from baseline after 48 weeks of treatment | Week 48
Proportion of subjects with weight loss of ≥15% from baseline after 48 weeks of treatment | Week 48
Change from baseline in waist circumference after 48 weeks of treatment | Baseline, Week 48
Change from baseline in weight after 48 weeks of treatment | Baseline, Week 48
Change from baseline in BMI after 48 weeks of treatment | Baseline, Week 48
Change from baseline in systolic blood pressure after 48 weeks of treatment | Baseline, Week 48
Change from baseline in diastolic blood pressure after 48 weeks of treatment | Baseline, Week 48
Change from baseline in Total Cholesterol after 48 weeks of treatment | Baseline, Week 48
Change from baseline in Low Density Lipoprotein (LDL) Cholesterol after 48 weeks of treatment | Baseline, Week 48
Change from baseline in Triglycerides after 48 weeks of treatment | Baseline, Week 48
Change from baseline in High Density Lipoprotein (HDL) Cholesterol after 48 weeks of treatment | Baseline, Week 48
Change from baseline in fasting plasma glucose (FPG) after 48 weeks of treatment | Baseline, Week 48
Change from baseline in glycosylated haemoglobin (HbA1c) after 48 weeks of treatment | Baseline, Week 48
Change from baseline in fasting serum insulin after 48 weeks of treatment | Baseline, Week 48
Change in scores of SF-36 V2 from baseline after 48 weeks of treatment | Baseline, Week 48
Number of AEs during the trial | week 0 to week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided